CLINICAL TRIAL: NCT06051851
Title: Penpulimab Combined With Anlotinib and Nab-paclitaxel Plus Gemcitabine (PAAG) as First-line Treatment for Advanced Metastatic Pancreatic Cancer: a Prospective, Multicenter, Single-arm, Phase 2 Study
Brief Title: Penpulimab Combined With Anlotinib and Nab-paclitaxel Plus Gemcitabine as First-line Treatment for Advanced Metastatic Pancreatic Cancer
Acronym: RCT-PAAG
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-289-01
Record Dates: First submitted 2023-09-18; First posted 2023-09-25 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-07

CONDITIONS: Pancreatic Adenocarcinoma Metastatic
Keywords: advanced metastatic pancreatic cancer; Chemotherapy; immunotherapy; Targeted Therapy
MeSH Terms: interventions — penpulimab; anlotinib; Taxes; Gemcitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trial group (Experimental): penpulimab in combination with anlotinib and AG regimen in the first-line treatment of advanced metastatic pancreatic cancer
  Interventions: Drug: Penpulimab; Drug: Anlotinib; Drug: Nab paclitaxel; Drug: Gemcitabine
- Control group (Active Comparator): AG regimen in the first-line treatment of advanced metastatic pancreatic cancer
  Interventions: Drug: Nab paclitaxel; Drug: Gemcitabine

INTERVENTIONS:
Drug: Penpulimab — Penpulimab 200mg IV D1
  1 cycle every 21 days
  Arms: Trial group
Drug: Anlotinib — Anlotinib 12mg/10mg P.O. QD D1-14 (12mg for body surface area ≥1.6m2, 10mg for body surface area ≤1.6m2)
  1 cycle every 21 days
  Arms: Trial group
Drug: Nab paclitaxel — Nab-paclitaxel 125mg/m2 I.V. D1,8
  1 cycle every 21 days
Drug: Gemcitabine — Gemcitabine 1.0g/m2 I.V. D1,8
  1 cycle every 21 days

SUMMARY:
This is a multi-center, open-label， randomized controlled Phase II clinical study to observe and evaluate the efficacy and safety of Penpulimab combined with Anlotinib and Nab-paclitaxel plus Gemcitabine (PAAG ) versus AG first-line treatment in patients with metastatic pancreatic cancer.

DETAILED DESCRIPTION:
This study is a multi-center, open-label, randomized controlled Phase II clinical study to evaluate the efficacy and safety of penpulimab in combination with anlotinib and AG regimen in the first-line treatment of advanced metastatic pancreatic cancer, and to explore the clinical indicators related to efficacy to guide the individualized treatment.

Trial group:

Nab-paclitaxel 125mg/m2 I.V. D1,8 Gemcitabine 1.0g/m2 I.V. D1,8 Penpulimab 200mg IV D1 Anlotinib 12mg/10mg P.O. QD D1-14 (12mg for body surface area ≥1.6m2, 10mg for body surface area ≤1.6m2)

Control group:

Nab-paclitaxel 125mg/m2 I.V. D1,8 Gemcitabine 1.0g/m2 I.V. D1,8

1 cycle every 21 days Efficacy assessments will be performed every 2 cycles for the first 8 cycles of treatment. If treatment exceeds 8 cycles (24 weeks) in the trial group, maintenance therapy with anlotinib + PD1 and efficacy assessment every 2 cycles; in the control group, efficacy assessment every 2 cycles. Patient with disease control (CR+PR+SD) and tolerable adverse events were continued on the drug until discontinuation of the drug if efficacy was evaluated as disease progression (PD), if an intolerable adverse event occurred, or if the investigator deemed it unsuitable for the patient to continue on the treatment.

Efficacy Indicators Primary endpoint: median progression-free survival (mPFS) Secondary endpoint: objective response rate (ORR), disease control rate (DCR), median overall survival (mOS), safety; potential biological indicators for predicting efficacy (tumor tissue NGS assay, ctDNA, mRNA, and various immune cytokines in peripheral blood, etc.)

Safety evaluation indexes:

Observe the presence or absence of clinical adverse events such as myelosuppression, nausea, vomiting, liver damage, skin reactions (e.g., rash), pneumonitis, hypertension, proteinuria, fatigue, and nausea, etc., which are graded according to NCI criteria.

ELIGIBILITY:
Inclusion Criteria:

* Ages ≥18 years，ECOG ≤ 2，Estimated survival time > 3 months
* Histologically or Cytologically confirmed metastatic pancreatic adenocarcinoma
* Based on Response Evaluation Criteria In Solid Tumors (RECIST1.1), there should be at least one measurable lesion
* Patients have never received systematical anti-cancer therapy
* Laboratory examination meets the following requirements:

White blood cell (WBC) ≥3.0×109/L; absolute neutrophil count (ANC) ≥1.5×109/L; Hemoglobin (HB) ≥90g/L; platelet count(PLT) ≥75×109/L; Total bilirubin (TBIL) ≤1.5× normal upper limit (ULN); Alanine aminotransferase (ALT) and Aspartate aminotransferase (AST)≤2.5×ULN, if accompanied by liver metastasis, ALT and AST≤5×ULN; Serum creatinine (Cr) ≤1×ULN or creatinine clearance (CCr)≥50ml/min;

* Doppler ultrasound evaluation: left ventricular ejection fraction (LVEF) > 50%
* Patients of childbearing age should take appropriate protective measures before enrollment and during the trial
* Volunteer to join the study, sign the informed consent, have good compliance, and cooperate with follow-up
* Ability to follow the study protocol and follow-up procedures.

Exclusion Criteria:

* Patients have ever received any systematical anti-cancer therapy in the past
* Patients who participated in other clinical trials in the past 4 weeks
* According to the investigator, patients who surgically available or potentially treatable(Patients who voluntarily give up surgical treatment can be enrolled after evaluation by the investigator)
* Patients with moderate ascites requiring drainage
* Patients with CNS metastases and/or carcinomatous meningitis
* Patients with history of other primary malignancies except: 1) complete remission before enrollment for at least 2 years and requiring no additional treatment during the study period; 2) Adequately treated non-melanoma skin cancer or lentiform malignancy with no evidence of disease recurrence; 3) Adequately treated carcinoma in situ with no evidence of disease recurrence;
* Patients with autoimmune disease or immune deficiency who are treated with immunosuppressive drugs
* Patients with bleeding tendency.
* Pregnant or lactating women.
* Drug abuse, clinical or psychological or social factors that impact informed consent or the conduct of the study
* Patients who may be allergic to PD-1 monoclonal antibody, anlotinib, albumin-bound paclitaxel and gemcitabine

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 177 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival（PFS） | up to 1 years
  Progression-free Survival (PFS) (median) was determined using the number of months measured from the initial date of treatment to the date of documented progression, or the date of death (in the absence of progression) of participants. Progression is defined using RECIST v1.1, as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | up to 1 years
  Objective response rate is defined as the percentage of subjects whose best response was complete response (CR) or partial response (PR) according to the Response Evaluation Criteria In Solid Tumors Criteria(RECIST v1.1)
Disease Control Rate (DCR) | up to 1 years
  Disease control rate is defined as the percentage of subjects whose best response was CR, PR or stable disease (SD) according to the RECIST v1.1
Overall Survival (OS) | up to 2 years
  Overall Survival (OS) (median) is determined using the number of months measured from the initial date of treatment to the recorded date of death of participants.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Du, Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (1):
- The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No